CLINICAL TRIAL: NCT00102440
Title: A Phase 3, Randomized, Multicenter Study Comparing the Safety and Efficacy of Oral Febuxostat Versus Allopurinol in Subjects With Gout
Brief Title: Febuxostat Versus Allopurinol Control Trial in Subjects With Gout
Acronym: FACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C02-010; U1111-1114-0184 (Registry Identifier: WHO)
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Gout
Keywords: uric Acid; xanthine oxidase; tophi; Drug Therapy
MeSH Terms: conditions — Gout | interventions — Febuxostat; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Febuxostat 80 mg QD (Experimental)
  Interventions: Drug: Febuxostat
- Febuxostat 120 mg QD (Experimental)
  Interventions: Drug: Febuxostat
- Allopurinol 300 mg QD (Active Comparator)
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Febuxostat — Febuxostat 80 mg, orally, once daily for up to 52 weeks.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 80 mg QD
Drug: Febuxostat — Febuxostat 120 mg, orally, once daily for up to 52 weeks.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 120 mg QD
Drug: Allopurinol — Allopurinol 300 mg, capsules, orally, once daily for up to 52 weeks.
  Arms: Allopurinol 300 mg QD

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of febuxostat, once daily (QD), versus allopurinol in subjects with gout.

DETAILED DESCRIPTION:
This was a randomized, controlled, double-blind study of 52 weeks duration. Subjects receiving prior urate-lowering therapy underwent a 2-week washout period prior to randomization. Subjects were then randomized to one of three treatment groups: febuxostat 80 milligram (mg), febuxostat 120 mg, or allopurinol 300 mg. Naproxen (250 mg twice daily) or colchicine (0.6 mg once daily) was provided for prophylaxis of acute gout flares during the washout period and the first 8 weeks of double-blind treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the preliminary criteria of the American Rheumatism Association for the classification of the acute arthritis of primary gout.
* Serum uric acid ≥ 8.0 milligrams per deciliter (mg/dL) at Baseline

Exclusion Criteria:

* Serum creatinine >1.5 mg/dL
* Calculated creatinine clearance of <50 milliliters per minutes (mL/min)
* Pregnancy or lactation;
* Concurrent therapy with urate lowering agents, azathioprine, 6-mercaptopurine, thiazide diuretics, or medications containing aspirin (>325 mg) or other salicylates;
* Body Mass Index (BMI) >50 kilogram per meter²(kg/m²);
* A history of xanthinuria, active liver disease, or hepatic dysfunction;
* A history of alcohol abuse or intake of 14 or more alcohol-containing drinks/week.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2002-07; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- [Result] Becker MA, Schumacher HR Jr, Wortmann RL, MacDonald PA, Eustace D, Palo WA, Streit J, Joseph-Ridge N. Febuxostat compared with allopurinol in patients with hyperuricemia and gout. N Engl J Med. 2005 Dec 8;353(23):2450-61. doi: 10.1056/NEJMoa050373. PMID 16339094
- [Result] Becker MA, MacDonald PA, Hunt BJ, Lademacher C, Joseph-Ridge N. Determinants of the clinical outcomes of gout during the first year of urate-lowering therapy. Nucleosides Nucleotides Nucleic Acids. 2008 Jun;27(6):585-91. doi: 10.1080/15257770802136032. PMID 18600509
- [Result] Wortmann RL, Macdonald PA, Hunt B, Jackson RL. Effect of prophylaxis on gout flares after the initiation of urate-lowering therapy: analysis of data from three phase III trials. Clin Ther. 2010 Dec;32(14):2386-97. doi: 10.1016/j.clinthera.2011.01.008. PMID 21353107
- [Result] Chohan S, Becker MA, MacDonald PA, Chefo S, Jackson RL. Women with gout: efficacy and safety of urate-lowering with febuxostat and allopurinol. Arthritis Care Res (Hoboken). 2012 Feb;64(2):256-61. doi: 10.1002/acr.20680. PMID 22052584
- See also: American College of Rheumatology — http://www.rheumatology.org/
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 112 investigative sites, 106 in the United States and 6 in Canada, from 11 July 2002 to 20 February 2004.
Pre-assignment Details: Subjects currently receiving urate-lowering therapy discontinued those urate-lowering therapies and initiated prophylactic medications before enrollment in once daily (QD) treatment groups.
Groups:
- Febuxostat 80 mg QD: Febuxostat 80 mg, orally, once daily for up to 52 weeks.
- Febuxostat 120 mg QD: Febuxostat 120 mg, orally, once daily for up to 52 weeks.
- Allopurinol 300 mg QD: Allopurinol 300 mg, orally, once daily for up to 52 weeks.
Period: Overall Study
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Started | 256 | 251 | 253
Completed | 168 | 153 | 187
Not Completed | 88 | 98 | 66
Not completed — Lost to Follow-up | 25 | 18 | 21
Not completed — Adverse Event | 16 | 23 | 8
Not completed — Gout Flare | 10 | 28 | 9
Not completed — Personal Reason(s) | 19 | 13 | 13
Not completed — Other | 11 | 14 | 14
Not completed — Protocol Violation | 7 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD | Total
Number analyzed (Participants) | 256 | 251 | 253 | 760
Age, Customized [Number; unit: subjects]
  <45 years | 75 | 71 | 84 | 230
  45 years to <65 years | 140 | 133 | 125 | 398
  ≥65 years | 41 | 47 | 44 | 132
Age Continuous [Mean (Standard Deviation); unit: years] | 51.8 (11.69) | 52.0 (12.12) | 51.6 (12.63) | 51.8 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 10 | 31
  Male | 243 | 243 | 243 | 729
Body Mass Index [Number; unit: subjects]
  <18.5 kilogram per meter² (kg/m²) | 0 | 0 | 0 | 0
  18.5 kg/m² to <25 kg/m² | 15 | 12 | 7 | 34
  25 kg/m² to <30 kg/m² | 75 | 87 | 89 | 251
  ≥30 kg/m² | 166 | 152 | 154 | 472
  missing | 0 | 0 | 3 | 3
Calculated Creatinine Clearance [Number; unit: subjects] — Calculated creatinine clearance based on the Cockcroft-Gault equation using ideal body weight.
  subjects
    <50 milliliters per minute (mL/min) | 13 | 8 | 13 | 34
    50 mL/min to <80 mL/min | 77 | 90 | 68 | 235
    80 mL/min to <120 mL/min | 138 | 130 | 140 | 408
    ≥120 mL/min | 28 | 23 | 29 | 80
    missing | 0 | 0 | 3 | 3
Presence of Primary Palpable Tophus [Number; unit: subjects]
  Yes | 52 | 53 | 46 | 151
  No, but other tophi present | 1 | 2 | 3 | 6
  No and no other tophi present | 203 | 196 | 204 | 603
Race/Ethnicity [Number; unit: subjects]
  White | 193 | 199 | 195 | 587
  Black or African American | 24 | 20 | 18 | 62
  Hispanic | 22 | 17 | 19 | 58
  Asian | 10 | 9 | 6 | 25
  Other | 7 | 6 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With the Last 3 Serum Urate Levels <6.0 Milligrams Per Deciliter (mg/dL)
Description: Each subject's serum urate at the last 3 visits determined the subject's response for the primary efficacy variable. A subject who prematurely discontinued without least 3 postbaseline serum urate levels was considered a nonresponder; if at least 3 serum urate were obtained postbaseline, those 3 visits were used. The last 3 visits used may have differed for each subject.
Time Frame: Last 3 Visits (up to 52 weeks)
Population: Analysis was performed on the intent-to-treat (ITT) subjects, which were defined as all randomized subjects who took at least 1 dose of study drug and who had a baseline serum urate ≥8.0 mg/dL.
Measure: Number; unit: Percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 255 | 250 | 251
Percentage of subjects | 53 | 62 | 21
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Non-Inferiority or Equivalence — Non-inferiority of febuxostat 80 mg to allopurinol was declared if the value of the lower bound of the 97.5% confidence interval is > -10%; Difference in percentage = 32, 97.5% CI [23.1 to 41.3]
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Non-Inferiority or Equivalence — Non-inferiority of febuxostat 120 mg to allopurinol was declared if the value of the lower bound of the 97.5% confidence interval is > -10%; Difference in percentage = 41, 97.5% CI [31.5 to 49.5]
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — Comparisons of each febuxostat dose to allopurinol were adjusted to control the overall 0.05 level of significance for superiority by using Hochberg's method for multiple comparisons
Statistical Analysis 4: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 3]
Statistical Analysis 5: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.072, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

2. Secondary Outcome: Percentage of Subjects With Serum Urate <6.0 mg/dL at Week 28 Visit
Description: Serum urate values were obtained at the Week 28 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Week 28 visit was summarized.
Time Frame: Week 28
Population: Analysis was performed on the ITT subjects, which were defined as all randomized subjects who took at least 1 dose of study drug and who had a baseline serum urate ≥8.0 mg/dL. Missing data were not imputed.
Measure: Number; unit: Percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 186 | 159 | 199
Percentage of subjects | 72 | 82 | 42
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.031, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

3. Secondary Outcome: Percentage of Subjects With Serum Urate <6.0 mg/dL at Week 52 Visit
Description: Serum urate values were obtained at the Week 52 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Week 52 visit was summarized.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 159 | 145 | 178
Percentage of subjects | 81 | 82 | 39
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.883, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

4. Secondary Outcome: Percentage of Subjects With Serum Urate <6.0 mg/dL at Final Visit
Description: The percentage of subjects whose serum urate was <6.0 mg/dL at the final visit was summarized. The final visit was the last visit at which a serum urate value was collected. The timing of the final visit may have differed for each subject.
Time Frame: Final Visit (up to 52 weeks)
Population: as for outcome 2
Measure: Number; unit: Percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 249 | 242 | 242
Percentage of subjects | 74 | 80 | 36
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.164, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

5. Secondary Outcome: Percent Change From Baseline in Serum Urate Levels at Week 28.
Description: Serum urate values were obtained at the Week 28 visit. The percent change in serum urate was calculated as [(week 28 - baseline levels/baseline)]*100 and summarized.
Time Frame: Baseline and Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 186 | 159 | 199
percent change from baseline | -46.3 (15.76) | -53.5 (18.20) | -34.8 (12.92)
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — P-values for pairwise comparisons are from contrast within the framework of the one-way ANOVA model with treatment as a factor. Statistical significance was determined at the 0.05 level without adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percent Change From Baseline in Serum Urate Levels at Week 52.
Description: Serum urate values were obtained at the Week 52 visit. The percent change in serum urate was calculated as [(week 52 - baseline levels/baseline)]*100 and summarized.
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 159 | 145 | 178
percent change from baseline | -47.7 (17.50) | -53.0 (19.31) | -34.8 (13.56)
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.006, ANOVA — [p-value comment as in outcome 5, analysis 1]

7. Secondary Outcome: Percent Change From Baseline in Serum Urate Levels at Final Visit
Description: The percent change in serum urate from baseline to the Final visit was calculated as [(Final Visit - baseline levels/baseline)]*100 and summarized. The Final visit was the last visit with a serum urate value. The timing of the final visit may have differed for each subject.
Time Frame: Baseline and Final Visit (up to 52 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 249 | 242 | 242
percent change from baseline | -44.7 (19.10) | -51.5 (19.91) | -33.0 (15.33)
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]

8. Secondary Outcome: Percent Change From Baseline in Tophus Size at Week 28, as Determined by Physical Measurement, in Subjects With a Palpable Primary Tophus at Screening.
Description: The percent change from baseline in primary tophus size as determined by physical measurement was calculated as [(Week 28 - baseline sizes)/baseline]*100 for the subset of subjects with a primary palpable tophus at the Screening Visit. If the primary tophus was no longer palpable at the Week 28 visit, the size was assumed to be zero.
Time Frame: Baseline and Week 28
Population: Analysis was performed on the ITT subjects, which were defined as all randomized subjects who took at least 1 dose of study drug, had a baseline serum urate ≥8.0 mg/dL, and had a palpable primary tophus measured at baseline. Missing data were not imputed.
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 36 | 28 | 33
percent change from baseline | -29.5 [-66.0 to 4.1] | -49.5 [-80.0 to -34.9] | -28.6 [-54.9 to 0.0]
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p > 0.999, Wilcoxon (Mann-Whitney) — P-values for pairwise comparisons are from the Wilcoxon rank-sum test. Statistical significance was determined at the 0.05 level without adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.011, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.024, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

9. Secondary Outcome: Percent Change From Baseline in Tophus Size at Week 52, as Determined by Physical Measurement, in Subjects With a Palpable Primary Tophus at Screening.
Description: The percent change from baseline in primary tophus size as determined by physical measurement was calculated as [(Week 52 - baseline sizes)/baseline]*100 for the subset of subjects with a primary palpable tophus at the Screening Visit. If the primary tophus was no longer palpable at the Week 52 visit, the size was assumed to be zero.
Time Frame: Baseline and Week 52
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 32 | 26 | 30
percent change from baseline | -83.4 [-100 to -15.6] | -65.5 [-85.5 to -38.9] | -49.7 [-96.0 to 0.0]
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.083, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.164, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.619, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

10. Secondary Outcome: Percent Change From Baseline in Tophus Size at Final Visit, as Determined by Physical Measurement, in Subjects With a Palpable Primary Tophus at Screening.
Description: Percent change in primary tophus size was calculated as [(Final Visit - baseline sizes)/baseline]*100 for the subset of subjects with a primary palpable tophus at Screening. If tophus was not palpable at Final visit, the size was assumed to be 0. The timing of the final visit may have differed for each subject.
Time Frame: Baseline and Final Visit (up to 52 weeks)
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 50 | 51 | 44
percent change from baseline | -51.7 [-100 to -8.3] | -43.8 [-83.0 to 0.0] | -39.6 [-65.0 to 1.5]
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.080, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.372, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.246, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

11. Secondary Outcome: Change From Baseline in Total Number of Tophi at Week 28 in Subjects With Palpable Tophi at Screening.
Description: The change from baseline at Week 28 in the total number of tophi per subject was calculated for the subset of subjects with palpable tophi at the Screening Visit. If the tophi were no longer palpable at the Week 28 visit, the total count was assumed to be zero.
Time Frame: Baseline and Week 28
Population: Analysis was performed on the ITT subjects, which were defined as all randomized subjects who took at least 1 dose of study drug, had a baseline serum urate ≥8.0 mg/dL, and had palpable tophi at baseline. Missing data were not imputed.
Measure: Median (Inter-Quartile Range); unit: number of tophi
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 38 | 30 | 37
number of tophi | 0.0 [0.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.674, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.320, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.411, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

12. Secondary Outcome: Change From Baseline in Total Number of Tophi at Week 52 in Subjects With Palpable Tophi at Screening.
Description: The change from baseline at Week 52 in the total number of tophi per subject was calculated for the subset of subjects with palpable tophi at the Screening Visit. If the tophi were no longer palpable at the Week 52 visit, the total count was assumed to be zero.
Time Frame: Baseline and Week 52
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: number of tophi
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 33 | 28 | 35
number of tophi | 0.0 [-1.0 to 0.0] | -1.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0]
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.507, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.188, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.362, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

13. Secondary Outcome: Change From Baseline in Total Number of Tophi at Final Visit in Subjects With Palpable Tophi at Screening.
Description: Change in number of tophi/subject calculated for the subset of subjects with palpable tophi at Screening. If the tophi were not palpable at the Final Visit, total count was assumed to be 0. The timing of the final visit may have differed for each subject.
Time Frame: Baseline and Final Visit (up to 52 weeks)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: number of tophi
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 52 | 53 | 47
number of tophi | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0]
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.657, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.444, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.719, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 8, analysis 1]

14. Secondary Outcome: Percentage of Subjects Requiring Treatment for Gout Flares Between Weeks 8 and 52.
Description: The percentage of subjects requiring treatment for a gout flare between Weeks 8 and 52 of the double-blind treatment period was summarized. A subject who reported more than 1 gout flare during this period was counted only once.
Time Frame: Weeks 8 through 52
Population: Analysis was performed on the ITT subjects who had at least one dose of study drug between Weeks 8 and 52.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Number analyzed (Participants) | 228 | 215 | 234
percentage of subjects | 64 | 70 | 64
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p > 0.999, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Allopurinol 300 mg QD; Test type: Superiority or Other; p = 0.229, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.266, Fisher Exact — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

ADVERSE EVENTS:
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol 300 mg QD
Serious Adverse Events (participants affected / at risk) | 10/256 | 19/251 | 18/253
Other Adverse Events (participants affected / at risk) | 164/256 | 145/251 | 167/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 80 mg QD (N=256) | Febuxostat 120 mg QD (N=251) | Allopurinol 300 mg QD (N=253)
Cardiac Disorders not elsewhere classified (NEC) (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Disorders NEC (Cardiac disorders) | 0 | 0 | 4
Heart Failures NEC (Cardiac disorders) | 3 | 1 | 0
Ischaemic Coronary Artery Disorders NEC (Cardiac disorders) | 3 | 2 | 2
Rate and Rhythm Disorders NEC (Cardiac disorders) | 0 | 0 | 1
Supraventricular Arrhythmias (Cardiac disorders) | 1 | 1 | 0
Ventricular Arrhythmias and Cardiac Arrest (Cardiac disorders) | 0 | 2 | 1
Acute and Chronic Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Fistulae (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Ulcers and Perforation, Site Unspecified (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Haemorrhages (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Ulcers and Perforation NEC (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal and Retroperitoneal Haemorrhages (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical Hernias (Gastrointestinal disorders) | 0 | 0 | 1
Febrile Disorders (General disorders) | 0 | 1 | 0
Allergies to Food, Food Additives, Drugs and Other Chemicals (Immune system disorders) | 1 | 0 | 0
Abdominal and Gastrointestinal Infections (Infections and infestations) | 0 | 1 | 2
Infections NEC (Infections and infestations) | 1 | 0 | 0
Lower Respiratory Tract and Lung Infections (Infections and infestations) | 0 | 1 | 0
Skin Structures and Soft Tissue Infections (Infections and infestations) | 0 | 1 | 0
Staphylococcal Infections (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infections (Infections and infestations) | 0 | 1 | 0
Viral Infections NEC (Infections and infestations) | 0 | 1 | 0
Chest and Lung Injuries NEC (Injury, poisoning and procedural complications) | 1 | 0 | 0
Non-Site Specific Injuries NEC (Injury, poisoning and procedural complications) | 1 | 0 | 0
Site Specific Injuries NEC (Injury, poisoning and procedural complications) | 1 | 0 | 0
Coagulation and Bleeding Analyses (Investigations) | 1 | 0 | 0
Joint Related Signs and Symptoms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal and Connective Tissue Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spine and Neck Deformities (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Colonic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostatic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Testicular Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Central Nervous System Vascular Disorders NEC (Nervous system disorders) | 0 | 1 | 0
Central nervous system Hemorrhages & Cerebrovascular Accidents (Nervous system disorders) | 0 | 1 | 0
Cervical Spinal Cord and Nerve Root Disorders (Nervous system disorders) | 0 | 1 | 0
Disturbances in Consciousness NEC (Nervous system disorders) | 0 | 1 | 1
Encephalopathies NEC (Nervous system disorders) | 0 | 1 | 0
Renal Failure and Impairment (Renal and urinary disorders) | 2 | 0 | 0
Renal Lithiasis (Renal and urinary disorders) | 0 | 0 | 1
Bronchospasm and Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax and Pleural Effusions NEC (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Thrombotic and Embolic Conditions (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failures (Excluding [Excl] Neonatal) (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Peripheral Embolism and Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 80 mg QD (N=256) | Febuxostat 120 mg QD (N=251) | Allopurinol 300 mg QD (N=253)
Diarrhoea (Excl Infective) (Gastrointestinal disorders) | 27 | 25 | 16
Nausea and Vomiting Symptoms (Gastrointestinal disorders) | 19 | 13 | 8
Oedema NEC (General disorders) | 18 | 8 | 8
Influenza Viral Infections (Infections and infestations) | 12 | 13 | 12
Lower Respiratory Tract and Lung Infections (Infections and infestations) | 13 | 7 | 8
Upper Respiratory Tract Infections (Infections and infestations) | 77 | 53 | 72
Limb Injuries NEC (Including [Incl] Traumatic Amputation) (Injury, poisoning and procedural complications) | 12 | 10 | 11
Non-Site Specific Injuries NEC (Injury, poisoning and procedural complications) | 11 | 10 | 12
Liver Function Analyses (Investigations) | 13 | 16 | 12
Joint Related Signs and Symptoms (Musculoskeletal and connective tissue disorders) | 39 | 32 | 37
Musculoskeletal and Connective Tissue Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 35 | 38 | 37
Headache NEC (Nervous system disorders) | 23 | 23 | 22
Neurological Signs and Symptoms NEC (Nervous system disorders) | 17 | 9 | 7
Upper Respiratory Tract Signs and Symptoms (Respiratory, thoracic and mediastinal disorders) | 13 | 10 | 17
Vascular Hypertensive Disorders NEC (Vascular disorders) | 7 | 10 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.